CLINICAL TRIAL: NCT02024009
Title: A Multi-centre Randomised Study of Induction Chemotherapy Followed by Capecitabine (+/-Nelfinavir) With High or Standard Dose Radiotherapy for Locally Advanced Non-metastatic Pancreatic Cancer
Brief Title: Systemic Therapy and Chemoradiation in Advanced Localised Pancreatic Cancer - 2
Acronym: SCALOP-2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Celgene (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: OCTO_063
Record Dates: First submitted 2013-12-23; First posted 2013-12-31 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2021-07

CONDITIONS: Pancreatic Neoplasms (Locally Advanced Non-metastatic)
Keywords: chemoradiotherapy; nelfinavir; abraxane; gemcitabine; radiotherapy; capecitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Nelfinavir; Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A (Experimental): 12 weeks (3 cycles) of induction Gemcitabine and Nab-paclitaxel (GEMABX) chemotherapy then 1 cycle of GEMABX* whilst radiotherapy (RT) planned then capecitabine (830mg/m2 oral bd) + Nelfinavir** + 50.4 Grays (Gy) in 28# (arm A closed on 26Feb2020 due to lack of efficacy of nelfinavir)
  *1 cycle GEMABX = 28 day cycle of intravenous Abraxane 125mg/m2 followed by gemcitabine 1000mg/m2 on day 1, 8 and 15.
  Interventions: Drug: nab-paclitaxel; Radiation: 50.4Gy in 28#; Drug: Nelfinavir; Drug: Capecitabine; Drug: Gemcitabine
- Arm B (Experimental): 12 weeks (3 cycles) of induction GEMABX chemotherapy then 1 cycle of GEMABX* whilst RT planned then capecitabine (830mg/m2 oral bd) + 50.4Gy in 28#
  *1 cycle GEMABX = 28 day cycle of intravenous Abraxane 125mg/m2 followed by gemcitabine 1000mg/m2 on day 1, 8 and 15.
  Interventions: Drug: nab-paclitaxel; Radiation: 50.4Gy in 28#; Drug: Capecitabine; Drug: Gemcitabine
- Arm C (Experimental): 12 weeks (3 cycles) of induction GEMABX chemotherapy then
  1 cycle of GEMABX* whilst RT planned then capecitabine (830mg/m2 oral bd) + Nelfinavir** + 60Gy in 30# (arm C closed on 26Feb2020 due to lack of efficacy of nelfinavir)
  *1 cycle GEMABX = 28 day cycle of intravenous Abraxane 125mg/m2 followed by gemcitabine 1000mg/m2 on day 1, 8 and 15
  Interventions: Drug: nab-paclitaxel; Radiation: 60Gy in 30#; Drug: Nelfinavir; Drug: Gemcitabine
- Arm D (Experimental): 12 weeks (3 cycles) of induction GEMABX chemotherapy then
  1 cycle of GEMABX* whilst RT planned then capecitabine (830mg/m2 oral bd) + 60Gy in 30#
  *1 cycle GEMABX = 28 day cycle of intravenous Abraxane 125mg/m2 followed by gemcitabine 1000mg/m2 on day 1, 8 and 15.
  Interventions: Drug: nab-paclitaxel; Radiation: 60Gy in 30#; Drug: Gemcitabine

INTERVENTIONS:
Drug: nab-paclitaxel — Abraxane is a proprietary solvent-free, protein-stabilized formulation of paclitaxel comprised of paclitaxel and human albumin in a noncrystalline amorphous state
  Other Names: Abraxane
Radiation: 60Gy in 30#
  Arms: Arm C; Arm D
Radiation: 50.4Gy in 28#
  Arms: Arm A; Arm B
Drug: Nelfinavir — VIRACEPT® (nelfinavir mesylate) is an inhibitor of the human immunodeficiency virus (HIV) protease.
  Other Names: Viracept
  Arms: Arm A; Arm C
Drug: Capecitabine — Given in combination with gemcitabine, known as GemCap.
  Arms: Arm A; Arm B
Drug: Gemcitabine — Gemcitabine is indicated for treatment of patients with locally advanced or metastatic adenocarcinoma of the pancreas. It is administered as an infusion
  Other Names: GEMZAR

SUMMARY:
This study will evaluate the role of increasing radiotherapy dose and addition of nelfinavir to chemoradiotherapy (CRT) in patients with inoperable pancreatic cancer that has not spread beyond the pancreas.

Currently in the United Kingdom (UK), either chemotherapy alone or chemotherapy followed by CRT can be used in the management of inoperable pancreatic cancer that has not spread. CRT consists of 25-30 radiotherapy treatments in combination with chemotherapy. Although this treatment is effective in controlling local symptoms and slowing down the pace of cancer, in most cases it is unable to shrink it enough to make it operable. Some of the reasons for this could be the lack of oxygen and lack of blood flow within the tumour making it resistant to the effects of CRT. This study will investigate whether increasing the dose of radiotherapy, or increasing the oxygen and blood supply to the tumour by giving nelfinavir, or a combination of both, can improve outcomes. We also want to know what the additional toxicities from such intensive approaches are.

All participants will initially receive 12 weeks of chemotherapy, and those with stable or responding disease will receive further study treatment. The treatment allocation, initially to one of the four options, but as of 26Feb2020, to one of two options, as outlined below will be done at random by computer and neither the doctor nor the patient can choose the treatment option. The process of randomisation ensures that all treatment arms are equally balanced in terms of patient and tumour characteristics, and to reduce the possibility of bias.

The study will consist of 2 stages. In the 1st stage we aimed to find the right dose of nelfinavir to combine with CRT, requiring 27 participants of whom up to 18 will receive nelfinavir together with CRT. The Maximum Tolerated Dose of nelfinavir for Stage 2 has been established as 1250mg bd based on the data of 4 patients in the Stage 1, 1250mg cohort. In the 2nd stage, we want to find out the benefits of this approach over and above standard treatments and therefore we will recruit the order of 168 participants and allocate 96 to 1 of the 4 following treatment arms (As from 26Feb2020, randomisation will continue into one of two arms):

Arm A: Nelfinavir together with CRT (arm A closed on 26Feb2020) Arm B: CRT (without nelfinavir) Arm C: Nelfinavir together with CRT (but using a higher than conventional dose of radiotherapy) (arm C closed on 26Feb2020) Arm D: CRT without nelfinavir (but using a higher than conventional dose of radiotherapy) Participants allocated to any of the two arms, following closure of Arms A & C on 26Feb2020, will receive one further cycle of chemotherapy prior to starting chemoradiotherapy (without nelfinavir). This is to allow time for radiotherapy planning.

Participants who are ineligible or refuse randomisation will be treated as per local standard but will remain in the study for follow up every 12 weeks. Their data will contribute to an Overall Survival (OS) analysis.

DETAILED DESCRIPTION:
Pancreatic cancer has a poor outcome. Approximately 8000 cases are diagnosed in the UK each year and approximately 8000 patients die from the disease [1]. 20% of the patients are operable at diagnosis, 30-40% have locally advanced inoperable disease [LANPC] and another 40-50% have metastatic disease. Patients with LANPC have a relatively better prognosis compared to patients with metastatic disease (median overall survival 10-12 months and 5-6 months respectively). Currently, treatment options for LANPC include:

1. Primary chemotherapy
2. Primary chemoradiation (CRT) followed by adjuvant chemotherapy
3. Induction chemotherapy followed by CRT

Studies investigating primary chemotherapy vs. primary CRT have reported overall survival between ten to 12 months and there are conflicting reports as to whether chemotherapy alone or primary CRT is superior [2, 3].

More recently, there has been a shift to using induction chemotherapy to pre-select patients who are suitable for CRT. The LAP07 trial [4] compared chemotherapy alone (gemcitabine with/without erlotinib) versus same chemotherapy for 4 months followed by consolidation capecitabine-based CRT. The study aimed to recruit over 700 patients but closed early on recommendation of IDMC following a planned interim analysis after 442 patients. This study failed to show superiority of consolidation CRT over continuing chemotherapy alone (median overall survival 15.2 months vs. 16.4 months, log rank p=0.8) but confirmed good tolerance of CRT in multi-institutional setting (Grade 3/4 gastro-intestinal toxicity 5.9%; Grade 3/4 neutropenia 3.1%) [4]. The investigators concluded that both chemotherapy alone and consolidation CRT are options for this group of patients and further trials should investigate intensifying both radiotherapy (RT) and chemotherapy strategies.

In the UK, the recently reported SCALOP trial randomised patients to gemcitabine or capecitabine based CRT following 4 months of induction GEMCAP chemotherapy [5]. 114 patients were recruited from 28 centres over 2 years, and 74 non-progressive patients were randomised to CRT. This study demonstrated UK's feasibility to recruit to CRT trials in pancreatic cancer and deliver high quality RT within a well-controlled Radiotherapy Trials Quality Assurance programme coordinated by the NCRI RTTQA Group. SCALOP suggested superiority of capecitabine-based CRT over gemcitabine based-CRT in terms of overall survival (median overall survival 15.2 vs. 13.4 months, HR 0.39, p=0.012) and treatment related Grade 3/4 toxicity (haematological 0% vs. 18%, p=0.008; non-haematological 12% vs. 26%, p=0·12). The outcome/toxicity in the cape-RT arm was very similar to that reported in LAP07 study, and capecitabine could now be considered as the preferred radio-sensitizer in the context of pancreatic CRT.

The importance of local control in LANPC Although LANPC and metastatic pancreatic cancer have been traditionally treated similarly with chemotherapy under the premise that this is largely a systemic disease, recent developments in molecular and genetic aspects of pancreatic cancer would suggest that this disease is heterogeneous with different genetic subtypes and the systemic nature of the disease can no longer be assumed. Studies have shown that nearly a third of patients with LANPC die as a result of local progression of their disease rather than systemic spread; the loss of Dpc4 gene has been correlated with systemic spread of the disease whereas patients with intact Dpc4 have local tumour predominance [6, 7]. Local progression occurs in more than half the cases after conventional CRT (SCALOP unpublished data) and one study has shown that local failure may be a predictor of early mortality (HR 2.15; p=0.0074, [8]). One meta-analysis of 4,394 patients suggests that one-third of initially unresectable tumours may become operable following neo-adjuvant therapy [9], and improving local control is likely to become more relevant in the face of improved systemic treatment like GEMABX (gemcitabine + nab-paclitaxel) and FOLFIRINOX, as patients are likely to live long enough to develop local symptoms.

Radiotherapy dose escalation It is widely accepted that adenocarcinoma is a radio-resistant tumour and radiation doses of less than 60-70Gy are unlikely to eradicate the disease. However current pancreatic CRT schedules (45-54Gy in 25-30 fractions) are limited by the tolerance dose of the surrounding organs at risk (OARs), i.e., small bowel, duodenum, stomach, liver and kidneys. Using current dose schedules, local failure occurs in 40-60% cases despite CRT [8, 10, 11] and <5% of patients show radiological or pathological complete response following treatment [9, 12].

A small retrospective study has shown that RT dose ≥ 54Gy was associated with a trend towards improved overall survival (11.3 mo. vs. 6.8 mo., p=0.089) [13]. Another Phase I dose intensification study explored the role of escalating dose per fraction, and a higher Biological Equivalent Dose (BED) of RT was delivered (dose escalated from 50 to 60 Gy in 25 fractions, concurrent with gemcitabine 1000mg/m2 weekly) [14]. The recommended phase II dose was 55Gy in 25 fractions, at which the DLT (Dose Limiting toxicity) probability was 0.24; of the 50 patients recruited to the study, the median OS was 14.8 months with a 2-year OS of 30%; 12 underwent resection (R0=10) with a median OS of 32 months in resected patients. The promising outcome and acceptable toxicity seen in this study suggests that role of RT dose escalation should be further investigated in a randomised trial.

Although concerns about safe radiation doses to the surrounding critical organs has previously discouraged dose escalation studies, modern day technical advancement with Intensity Modulated radiotherapy (IMRT) and Image Guided RT (IGRT) allows precise delivery of radiotherapy while reducing dose to OARs [14-16]. A dose of 59.4Gy/33 fractions has been safely delivered in combination with gemcitabine, cisplatin and RT in the ARC I and the ARC II studies [17](see below ). A hypothetical planning study from the MD Anderson group has demonstrated that dose to the pancreas can be escalated to 72Gy/36 fractions based on relationship of GTV to the gastro intestinal-OARs, using IMRT or proton therapy [18]. Taken together, these studies indicate that radiation dose in the region of 60Gy using conventional fractionation and conservative radiation volumes could be investigated as a component of dose escalation in a multi-centre 'trial, within constraints of a rigorous Radiotherapy Quality Assurance programme.

Nelfinavir in pancreatic cancer CRT Pancreatic cancer remains refractory to most conventional therapies and is driven by multiple oncogenic mutations including KRAS mutation and PTEN loss. EGFR (Epidermal Growth Factor Receptor), KRAS and PIK3CA signalling are mediated in part through PI3K (Phospho-Inositol-3 Kinase) and Akt signalling. Preclinical data suggest that PI3K-inhibition using HIV protease inhibitors including nelfinavir reduce radioresistance [19, 20] and downregulates phosphorylation of Akt at Ser473 leading to radiosensitization [21, 22]. As Akt pathway is overactive in tumours but not normal tissue, it causes selective radiosensitization without aggravating RT mediated normal tissue damage. This radiosensitization effect is seen even in KRAS mutant pancreatic cell lines [19], which is highly relevant in clinical practice as >90% of pancreatic tumours are KRAS mutant. The inhibition of this pathway has also been shown to normalise tumour vasculature, increase vascular flow and perfusion and reduce hypoxia in tumour xenografts [23, 24], all of which may also contribute to the radiosensitizing effect seen with this class of drugs. As nelfinavir has been widely used as an anti-retroviral agent, there is a wealth of safety data on this agent [25] and a retrospective study has shown no increase in radiation related acute toxicity compared to control [26]. The ARC-I trial, a phase I study which tested the toxicity of nelfinavir-based CRT in LANPC. Twelve patients were treated with a RT dose of 59.4Gy radiation in 33 fractions in combination with nelfinavir (1250mg bd, starting 3 days before start of RT, until final day of RT), gemcitabine (Dose level 1: 200mg/m2; Dose level 2: 300mg/m2) and cisplatin 30mg/m2 with the chemotherapy being delivered on days 1, 8, 22, 29 [17]. Grade 3 /4 non-haematological toxicity was reported in 16.7%; complete radiological response on FDG-PET was seen in 50% of the cases and R0 resection was achieved in 6 patients. Median OS was 18 months. A subsequent phase II study, ARC II (35), tested the efficacy and toxicity of the combination at the higher dose of Gemcitabine (300mg/m2) in 23 patients. Although upfront CRT (without induction chemotherapy) was used, median and 1-year overall survival were 17.4 months and 73.4% respectively, which compares well historic studies of primary CRT. Key Grade 3/4 toxicities (nausea/vomiting 21.7%; diarrhoea 21.7%; fatigue 17.4%; neutropenia 8.7%; thrombocytopenia 39.1%) is likely to have been contributed by the gemcitabine/cisplatin chemotherapy and large RT fields which included prophylactic nodal irradiation. In addition to this study, a recently reported phase I study combining radical CRT with nelfinavir in stage IIIA and B non-small cell lung cancer showed minimal toxicity with five out of nine complete responses [27]. Nelfinavir has demonstrated promising radio-sensitizing effects and therefore merits further investigation in a phase II trial.

Systemic therapy in pancreatic cancer Both FOLFIRINOX (5FU, Folinic Acid, Irinotecan, Oxaliplatin) [28] and GEMABX [29] are treatment options for patients with good performance status advanced pancreatic cancer.

The MPACT study [29] compared gemcitabine alone with a combination of gemcitabine and nab-paclitaxel in 861 patients with metastatic pancreatic cancer. The OS (8.5 vs. 6.7 months, p<0.001), PFS (5.5 vs. 3.7 months, p<0.001) and overall response rate (23% vs. 7%, p<0.001) favoured the combination therapy. Although Grade 3/4 neutropenia was seen in 38% of patients (cf 27% on gemcitabine alone), incidence of febrile neutropenia was low (3%) and other toxicities were manageable (Grade 3/4 fatigue 17% vs. 7%; Grade 3/4 neuropathy 17% vs. 1%, improved to Grade 0/1 in 29 days). Relative protocol doses of gemcitabine and nab-paclitaxel were 75% and 81% respectively (cf 85% in the gemcitabine arm) and suggested that the regimen is well tolerated. Moreover, the relative lack of non-overlapping toxicity with capecitabine-RT, most importantly gastro-intestinal toxicity, makes it an attractive regimen to use prior to consolidation CRT.

2.3 Rationale Local control is important in pancreatic cancer but current CRT schedules could be refined. Improving local control through RT dose escalation or enhanced radiosensitization may improve local control and overall survival in pancreatic cancer. We wish to test this hypothesis in the SCALOP-2 trial.

ELIGIBILITY:
Inclusion criteria:

1. 1. Aged 18 years or over
2. Histologically or cytologically proven carcinoma of the pancreas
3. Locally advanced, non-metastatic inoperable disease as per NCCN criteria (APPENDIX 2). The following types of interventions are allowed:

   1. Palliative bypass procedure
   2. Common bile duct stenting
4. Primary pancreatic lesion 6 cm or less in diameter (taken from scan results)
5. World Health Organisation PS 0-1 (APPENDIX 1)
6. Adequate haematological function: neutrophils ≥1.5 x 109/L, platelets ≥100 x 109/L
7. Adequate liver function tests:

   1. Serum bilirubin ≤1.5 x ULN. In participants who have had a recent biliary drain and whose bilirubin is improving, a value of ≤3 x ULN is acceptable, however treatment should not start unless Bilirubin is ≤1.5 x ULN.
   2. AST and/or ALT ≤ 3 x ULN.
8. Adequate renal function (GFR ≥ 40ml/min (Cockcroft & Gault - APPENDIX 3))
9. Written informed consent obtained
10. Women of child-bearing potential (APPENDIX 6) must have negative serum or urine pregnancy test within 14 days prior to registration, must agree to use a highly effective contraception method during GEMABX treatment and for 6 months after last administration of GEMABX and to use an acceptable contraception method during chemoradiotherapy and for 6 months after completion of all treatment. (For a definition of highly effective and acceptable contraceptive methods see section 10.8)
11. Male patients must be surgically sterile or must agree to use a condom during GEMABX treatment and for 6 months after last administration of GEMABX, and to use a condom during chemoradiotherapy and for three months after completion of chemoradiotherapy or, whichever date comes last.

Exclusion criteria:

1. Primary resectable cancer of the pancreas.
2. Distant metastases
3. Pregnant or breast-feeding patients.
4. Any evidence of severe uncontrolled systemic diseases including uncontrolled coronary artery disease, myocardial infarction or stroke within the last 6 months, any major systemic or psychiatric co-morbidities or any other considerations that the PI judges might impact on patient safety or protocol compliance and achievement of the study aims.
5. Previous malignancies in the preceding 3 years except for:

   1. In situ cancer of the uterine cervix
   2. Adequately treated basal cell skin carcinoma
   3. Adequately treated early stage non-pancreatic malignancy in complete remission for at least 3 years
6. Renal abnormalities including adult polycystic kidney disease or hydronephrosis or ipsilateral single kidney (i.e. functioning right kidney for head tumours; left kidney for tail tumours) that may preclude upper abdominal radiotherapy without damaging functional kidneys.
7. Previous RT to upper abdomen
8. Recurrent cancer following definitive pancreatic surgery
9. Lymphoma or neuroendocrine tumours of the pancreas
10. Known haemophilia A and B, chronic hepatitis type B or C.
11. Other experimental treatment 6 weeks or less prior to registration into this study (including chemothera¬py and immunotherapy).
12. Known hypersensitivity to any of the IMPs or any of their excipients.
13. Known dihydropyrimidine dehydrogenase (DPD) deficiency
14. Known galactose intolerance, Lapp-lactose deficiency or glucose-galactose malabsorption
15. History of severe unexpected reaction to fluoropyrimidine therapies
16. If the following concomitant medications cannot be discontinued temporarily during the CRT phase then the patients cannot enter the trial as they interact with capecitabine:

    1. Sorivudine and analogues e.g. brivudine
    2. Methotrexate.
    3. Allopurinol and dipyridamole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Progression free survival | From date of registration until date of first documented progression or death ( if death occurred without progression), assessed up until last patient last visit (43 months).
  Concurrent biological question (± Nelfinavir): Progression Free Survival (PFS) (time from registration to event (progression or death if death occurred without progression). Patients who are not assessed to have disease progression and are not observed to die during the course of the trial will be censored at the last known progression free follow-up date).
Overall survival in LANPC | From date of registration until date of first documented (death by any cause), assessed up until Last Patient Last Visit (43 months)
  RT dose question (50.4Gy v 60Gy): Overall survival (OS) (time from registration to event (death by any cause); patients who are not observed to die during the course of the trial will be censored at the last known date alive prior to end of trial date)

SECONDARY OUTCOMES:
Concurrent biological question: Toxicity (Serious Adverse Events scored by using NCI CTCAE v4.03), | 12 months from date of registration
  Toxicity (-nelfinavir vs. +nelfinavir; 50.4Gy vs. 60Gy): Serious Adverse Events will be scored using the NCI CTCAE v4.03 at registration, during treatment, post treatment and during follow up of randomised participants. Serious adverse events will be collected in "real-time".
Concurrent biological question: treatment compliance measured using patient diary cards | 12 months from date of registration
  Chemotherapy treatment compliance (-nelfinavir vs. +nelfinavir) measured through use of patient diary cards to count the number of days patient indicated they had taken the prescribed dose.
Concurrent biological question: overall survival | 12 months from date of registration
  -Overall survival: (-nelfinavir vs. +nelfinavir): Time from registration to death by any cause and those still alive will be censored at time last known alive
Concurrent biological question: resection rates | 12 months from date of registration
  -Resection rates: • Surgical resection (of primary tumour) rate (-nelfinavir vs. +nelfinavir; 50.4Gy vs. 60Gy)
RT dose question: PFS | 12 months from date of registration
  • Progression free survival (time to event (progression)) (50.4Gy vs. 60Gy) ,
RT dose question: 12-month OS rate, | 12 months from date of registration
  • Progression free survival (time to event (progression)) (50.4Gy vs. 60Gy) ,
RT dose question: resection rates, | 12 months from date of registration
  • Progression free survival (time to event (progression)) (50.4Gy vs. 60Gy) ,
Quality of life assessment by EORTC QLQ-C30 questionnaire | Quality of life using EORTC QLQ-C30 questionnaire was assessed at baseline, month 4 , 8 30, 39, 52 .
  Quality of life will be assessed by the EORTC QLQ-C30 V3.0 scoring system which uses the participant response categories "Not at all, "A little", "Quite a bit" and "Very much" to 30 questions on heath.
Quality of life assessment by PAN26 questionnaire | Quality of life using PAN26 questionnaire was assessed at baseline, month 4 , 8 30, 39, 52 .
  Quality of life will be assessed by the PAN26 V1.0 scoring system which uses the participant response categories "Not at all, "A little", "Quite a bit" and "Very much" to 25 questions on health-related symptoms and problems.
Quality of life assessment by the EQ-5D questionnaire | Quality of life using the EQ-5D questionnaire was assessed at baseline, month 4 , 8 30, 39, 52 .
  Quality of life will be assessed by the EQ-5D questionnaire V1.0 using 5 categories of health related questions asking participants to identify which sentence best describes them from" I have no problems to..." until "I am unable to...."and a scale from 0-100 (100 means the best health you can imagine, 0 means the worst health you can imagine).
CA19-9 level, 1-year local control rate | 12 months from date of registration
  • CA19-9 level: in units per ml
Disease response | 12 months from date of registration
  Disease response at each CT scan based on RECIST v1.1 in APPENDIX 4: complete response, partial response, progressive disease, stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Somnath Mukherjee, MD, FRCP, FRCR, Principal Investigator — somnath.mukherjee@oncology.ox.ac.uk
Locations (23):
- United Kingdom (23):
  - Oxford University Hospitals, Churchill Cancer Centre, Headington, Oxfordshire
  - NHS Grampian, Aberdeen Royal Infirmary, Aberdeen
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington
  - Belfast Health and Social Care Trust, Belfast City Hospital, Belfast
  - University Hospitals Bristol NHS Foundation Trust, Bristol Haematology and Oncology Centre, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Addenbrooke's Hospital, Cambridge
  - Velindre NHS Trust, Velindre Cancer Centre, Cardiff
  - East Suffolk and North Essex NHS Foundation Trust, Colchester District General Hospital, Colchester
  - Hull and East Yorkshire Hospitals NHS Trust, Castle Hill Hospital, Cottingham
  - University Hospitals Coventry and Warwickshire NHS Trust, University Hospital Coventry, Coventry
  - Royal Surrey County Hospital, Guildford
  - Leeds Teaching Hospitals NHS Trust, St James's University Hospital, Leeds
  - United Lincolnshire Hospitals NHS Trust, Lincoln County Hospital, Lincoln
  - North Middlesex University Hospital NHS Trust, North Middlesex Hospital, London
  - University College London Hospitals NHS Foundation Trust, University College London Hospital, London
  - Royal Free Hampstead NHS Trust, Royal Free Hospital, London
  - Hammersmith Hospital, London
  - The Christie NHS Foundation Trust, The Christie Hospital, Manchester
  - Milton Keynes University Hospital, Milton Keynes
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham University Hospitals NHS Trust, City Hospital, Nottingham
  - Plymouth Hospitals NHS Trust, Derriford Hospital, Plymouth
  - Sheffield Teaching Hospitals, Weston Park Hospital, Sheffield

REFERENCES:
- [Derived] Strauss VY, Shaw R, Virdee PS, Hurt CN, Ward E, Tranter B, Patel N, Bridgewater J, Parsons P, Radhakrishna G, O'Neill E, Sebag-Montefiore D, Hawkins M, Corrie PG, Maughan T, Mukherjee S. Study protocol: a multi-centre randomised study of induction chemotherapy followed by capecitabine +/- nelfinavir with high- or standard-dose radiotherapy for locally advanced pancreatic cancer (SCALOP-2). BMC Cancer. 2019 Feb 4;19(1):121. doi: 10.1186/s12885-019-5307-z. PMID 30717707